CLINICAL TRIAL: NCT03628833
Title: Hill-Rom Incontinence Management System ICU Field Evaluation
Brief Title: Incontinence Management System ICU Field Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-CWS2018-002
Record Dates: First submitted 2018-07-09; First posted 2018-08-14 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-08

CONDITIONS: Urinary Incontinence; Fecal Incontinence
MeSH Terms: conditions — Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Incontinence Management system (Experimental)
  Interventions: Device: Incontinence Management System

INTERVENTIONS:
Device: Incontinence Management System — Incontinence detection device

SUMMARY:
The objective of this Field Evaluation is to assess usage and satisfaction associated with the Hill-Rom Incontinence Management System.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urinary, fecal, or dual incontinence who are ≥ 18 years old
* The patient, or the patient's legal authorized representative (LAR), is willing and able to provide written informed consent

Exclusion Criteria:

- Patients that are considered to be near death or require palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Staff satisfaction surveys on product performance | Through study completion, an average of 4 months
  Following product use, staff can complete an optional, Likert scale survey

SECONDARY OUTCOMES:
Patient exposure time following an incontinence event | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No